CLINICAL TRIAL: NCT07232095
Title: 7-Day Vonoprazan-High-Dose Amoxicillin-Bismuth Therapy for First-Line Eradication of Helicobacter Pylori: A Multicenter Randomized Controlled Trial
Brief Title: 7-Day Vonoprazan, High-Dose Amoxicillin, and Bismuth Therapy
Acronym: JSHERO4
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Ye, Associate professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025JSHERO4
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter Pylori; Vonoprazan; Amoxicillin; Bismuth; Eradication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-day Vonoprazan-High-dose Amoxicillin-Bismuth therapy (Experimental): Vonoprazan 20mg twice daily+Amoxicillin 1g three times daily+Bismuth 220mg twice daily for 7 days
  Interventions: Drug: VAB-7
- 14-day Vonoprazan-Amoxicillin dual therapy (Active Comparator): Vonoprazan 20mg twice daily and Amoxicillin 1g three times daily for 14 days
  Interventions: Drug: VA-14

INTERVENTIONS:
Drug: VAB-7 — Vonoprazan 20mg twice daily+Amoxicillin 1g three times daily+Bismuth 220mg twice daily for 7 days
  Arms: 7-day Vonoprazan-High-dose Amoxicillin-Bismuth therapy
Drug: VA-14 — Vonoprazan 20mg twice daily and Amoxicillin 1g three times daily for 14 days
  Arms: 14-day Vonoprazan-Amoxicillin dual therapy

SUMMARY:
The 2024 American College of Gastroenterology (ACG) Clinical Guideline recommends a 14-day vonoprazan-amoxicillin (VA) regimen, consisting of vonoprazan 20 mg twice daily with amoxicillin 1000 mg three times daily, as a first-line treatment for Helicobacter pylori (H. pylori) infection.

Our previous study on regimen optimization showed that vonoprazan 20 mg twice daily combined with amoxicillin 1 g three times daily or 750 mg four times daily for 10 days achieved satisfactory eradication rates exceeding 90%, with no significant difference between dosing frequencies. However, when the treatment duration was shortened to 7 days, both dosing schedules failed to reach satisfactory eradication rates, indicating a need for further optimization.

Bismuth has antibacterial and synergistic properties, such as disrupting bacterial membranes, suppressing protein synthesis, and reducing virulence factor expression. It may enhance the efficacy of antibiotics. Therefore, this study evaluated the efficacy and safety of a 7-day vonoprazan-high-dose amoxicillin-bismuth (VAB-7) regimen as a first-line treatment for H. pylori infection.

Eligible participants in this study will be randomly assigned to one of the following treatment groups based on a pre-generated randomization sequence:

Control Group: Vonoprazan combined with high-dose amoxicillin dual therapy for 14 days (VA-14): Vonoprazan 20mg twice daily + Amoxicillin 1g three times daily.

Experimental Group: Vonoprazan combined with high-dose amoxicillin and bismuth therapy for 7 days (VAB-7): Vonoprazan 20mg twice daily + Amoxicillin 1g three times daily+Bismuth 220mg twice daily.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a Gram-negative bacterium that chronically colonizes the gastric mucosa, leading to persistent inflammation and mucosal injury. Eradication of H. pylori can prevent the recurrence of peptic ulcers, treat gastric mucosa-associated lymphoid tissue (MALT) lymphoma, and reduce the risk of gastric cancer. However, with the increasing prevalence of antibiotic resistance, eradication rates have gradually declined worldwide, creating an urgent need for more effective, safe, and practical treatment regimens.

In recent years, vonoprazan, a novel and potent potassium-competitive acid blocker (P-CAB), has emerged as an alternative to conventional proton pump inhibitors (PPIs). Its rapid onset and strong acid suppression provide an ideal environment for amoxicillin to maintain stable bactericidal activity. The vonoprazan-amoxicillin (VA) dual therapy has demonstrated excellent eradication efficacy and safety in several clinical studies and has been recommended by the 2024 American College of Gastroenterology (ACG) Clinical Guideline as a first-line treatment for H. pylori infection.

Our previous multicenter trial on regimen optimization showed that vonoprazan 20 mg twice daily combined with amoxicillin 1 g three times daily or 750 mg four times daily for 10 days achieved satisfactory eradication rates above 90%, with no significant difference between dosing frequencies. However, shortening the treatment duration to 7 days resulted in slightly lower eradication rates (below 90%), indicating that the shortened regimen may require further optimization to maintain high efficacy.

Bismuth compounds exhibit multiple antimicrobial and synergistic effects. They can inhibit H. pylori adhesion to the gastric mucosa, disrupt bacterial membrane integrity, suppress protein synthesis, and reduce the expression of virulence factors. In addition, bismuth enhances the activity of antibiotics such as amoxicillin by reducing bacterial resistance and increasing local drug concentration in the gastric mucosa. Previous studies have shown that 7-day bismuth-containing regimens(with amoxicillin and tetracycline) can achieve comparable eradication rates to 14-day regimens.

This study was designed to evaluate whether the addition of bismuth could improve the efficacy of a short-course vonoprazan-amoxicillin regimen. Specifically, the trial investigates the 7-day vonoprazan-high-dose amoxicillin-bismuth (VAB-7) regimen as a first-line treatment for H. pylori infection.

This multicenter, randomized, controlled trial aims to compare the efficacy and safety of VAB-7 with the standard 14-day vonoprazan-high-dose amoxicillin dual therapy (VA-14). The primary endpoint is the eradication rate of H. pylori confirmed by a ¹³C-urea breath test performed at least 4 weeks after treatment completion. Secondary outcomes include adverse event rates, patient adherence, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years, regardless of sex.
2. Helicobacter pylori infection confirmed by ¹³C or ¹⁴C urea breath test within 1 month before enrollment.
3. Chronic gastritis with H. pylori infection confirmed by endoscopy within 3 months, meeting the indications for eradication therapy in the Sixth National Consensus Report on the Management of Helicobacter pylori Infection (China), and willing to receive eradication treatment.
4. No prior H. pylori eradication therapy.
5. Written informed consent before participation.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any study medication (vonoprazan, amoxicillin, or bismuth).
2. Use of potassium-competitive acid blockers (P-CABs), proton pump inhibitors (PPIs), H₂ receptor antagonists, antibiotics, bismuth preparations, or probiotics within 4 weeks before enrollment.
3. Pregnant or lactating women.
4. Concomitant use of nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroids, or anticoagulants during the study period.
5. Presence of serious comorbid conditions that may interfere with study evaluation, including significant cardiac, pulmonary, hepatic, renal, metabolic, or psychiatric disorders, or malignancy.
6. History of gastric or esophageal surgery.
7. Any condition or factor that may affect compliance or make it difficult for the subject to complete follow-up as required.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 4-6 weeks after treatment completion
  Rate of H. pylori successfully eradicated; The confirmation of H. pylori status was evaluated by Urea breath test.

SECONDARY OUTCOMES:
Patient compliance | 1 day after treatment completion
  Good compliance was defined as achieving ≥80% of drugs in the regimes and bad compliance was defined as achieving <80% of drugs.
Adverse events | For the 7-day intervention: assessment on Day 3 and Day 7; For the 14-day intervention: assessment on Day 7 and Day 14.
  Adverse drug reactions, including the incidence of both overall and serious adverse events, will be assessed using a standardized questionnaire.
Cost-effectiveness ratio | 1 day after the procedure
  The cost-effectiveness ratio is defined as the total cost per patient for one course of H. pylori eradication treatment divided by the H. pylori eradication rate.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No